CLINICAL TRIAL: NCT06402214
Title: The 'Lombard Effect' in Patients Affected by Adductor Laryngeal Dystonia: a Pilot Study
Brief Title: The 'Lombard Effect' in Patients Affected by Adductor Laryngeal Dystonia
Acronym: LoQVAdSD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ID 6117
Record Dates: First submitted 2024-04-19; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Adductor Spasmodic Dysphonia
Keywords: laryngeal dystonia; spasmodic dysphonia; Lombard effect; auditory system
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Experimental): patients affected by adductor laryngeal dystonia
  Interventions: Other: Lombard test
- Control group (Active Comparator): healthy patients
  Interventions: Other: Lombard test

INTERVENTIONS:
Other: Lombard test — In this study a single-subject enrolment session will be set up, with the presence of a dedicated physician for informed consent, the performance of a tonal audiometric examination and a clinical practice phoniatric examination for all enrolled subjects, the collection of voice recordings both before and during the Lombard Test (LT) and the administration of the rating scales both before and after the LT performance. For each subject, voice recordings will be made of the vowel /a/ sustained for at least four seconds with a comfortable tone and volume and of the speech obtained from the reading aloud and volume of normal conversation of a phonetically balanced text (The Desert) lasting about 1 minute, first in a silent condition and then in the presence of noise. Specifically, for the LT, each subject will be exposed to a free-fieldwhite noise of speech(SWN) administered through headphones. The intensity of the noise will be 70 dB SPL. Voice recordings will be made in a quiet room.

SUMMARY:
Adductory spasmodic dysphonia (AdSD) is a rare condition characterised by irregular and uncontrolled voice interruptions, most commonly affecting women around the age of 45. The diagnosis is clinical and usually requires evaluation by several specialists. The exact cause is not known, but a disturbance of the motor system is hypothesised, probably related to various causes such as loss of cortical inhibition or problems with sensory input.

Neuroimaging studies have shown hyperactivity in various brain regions during speech production in patients with AdSD, but it is still unclear whether this hyperactivity is due to a malfunction of auditory and somatosensory feedback or an impairment of motor programming.

Recent research indicates that patients with AdSD show excessive muscle activation during phonation, probably due to abnormal processing of auditory feedback. This suggests that intervention in the auditory system may offer new treatment opportunities.

The proposed study aims to describe the acoustic, auditory-perceptual and subjective voice and speech changes in AdSD subjects during the Quick-Lombard Test (LT), a test that assesses vocal response under noisy conditions.

ELIGIBILITY:
Inclusion Criteria:

* Native Italian-speaking patients;
* Normal hearing, hearing threshold < 20 dB HL for frequencies from 0.5 to 4 KHz;
* Age >18 years and <65 years;
* Written informed consent.

Exclusion Criteria:

* Non-Italian-speaking patients.
* Patients undergoing treatment for dystonia.
* Previous laryngeal surgery.
* Patient undergoing speech therapy.
* Patient undergoing dopaminergic therapy.
* Inability to sustain phonation of sufficient duration >3 seconds or to perform sufficient tests to assess vocal outcomes.
* Lack of written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
OMNI Vocal Effort Scale | At the time of enrollement
  It is a validated instrument for the assessment of vocal effort perceived by the patient with AdSD. The OMNI-VES is a visual analogue scale 0-10 with graphic representation of vocal effort. The OMNI-VES will be administered under silent conditions and after the LT
Auditory-perceptual assessment | At the time of enrollement
  Blinded perceptual assessment, using the Global Grading Scale - Hoarseness - Straining - Asthenia - Straining (GRBAS) 0-3 (0 = normal; 1 = mild; 2 = moderate; 3 = severe) will be performed on the recorded voice samples by two speech therapists who will not be involved in the patients' care. Each voice sample will be anonymised and randomly distributed to the assessors.
Maximum Phonation Time | at the time of enrollement
  The maximum phonatory time (TMF) will be obtained by asking the subject to sustain the vowel /a/ as long as possible in one breath. The longest of the three attempts will be calculated as TMF in seconds. The TMF will be obtained before and during LT.
Average Frequency (Hz) | At the time of enrollement
  The Average Frequency is the fundamental frequency of the voice (pitch) usually ranges from approximately 30-300 Hz, but this varies according to different speakers: typically males' pitch ranges from 50-180Hz and females from 80-250Hz, so we usually set the pitch range to a reasonable range of 50-400Hz for general usage
Maximum Frequency (Hz) | At the time of enrollement
  The Maximum Frequency (Hz) is the highest frequency recorded within the voice signal
Maximum Intensity (dB SPL) | At the time of enrollement
  The Maximum Intensity (dB SPL) parameter refers to the highest intensity of the recorded voice signal
Degree of Voice Interruptions (%) | At the time of enrollement
  Degree of Voice Interruptions (%) is useful for the evaluation of temporary vocal interruption
Cepstral Peak Prominence-Smoothed (CPPS) | At the time of enrollement
  Cepstral Peak Prominence-Smoothed (CPPS) has been defined as a spectrum of a spectrum, whereby an inverse Fast Fourier Transform of the natural log of a frequency-domain spectrum is applied, transforming the spectrum to the time domain. The cepstral peak (CP) is a representation of the most dominant peak in the cepstrum - normally the fundamental frequency (fo) in a type I signal. After its first applications to voice was established the method of normalizing the amplitude of the overall cepstrum using a linear regression line. When applied to the cepstrum, the level difference (dB) between the cepstral peak and the regression line at the same quefrency provides the cepstral peak prominence (CPP). The CPPS values obtained from speech and vowel tasks proved reliable in predicting overall grade of dysphonia as well as breathiness.
Number of Voice Interruptions | At the time of enrollement
  Number of Voice Interruptions is useful for the evaluation of temporary vocal interruption

CONTACTS AND LOCATIONS:
Overall Officials: Maria Raffaella Marchese, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No
The data are paper-based